CLINICAL TRIAL: NCT02652468
Title: A Pilot Study to Assess Engraftment Using CliniMACS TCR-α/β and CD19 Depleted Stem Cell Grafts From Haploidentical Donors for Hematopoietic Progenitor Cell Transplantation (HSCT) in Patients With Relapsed Lymphoma
Brief Title: TCR-α/β and CD19 Depleted Stem Cell Grafts From Haplo Donors for HSCT in Relapsed Lymphoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW14113; 2015-0996 (Other: IRB); NCI-2015-02269 (Registry Identifier: NCI Trial ID); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison); Protocol Version 4/24/2020 (Other: UW Madison)
Record Dates: First submitted 2016-01-05; First posted 2016-01-11 (Estimated); Results first posted 2020-01-13 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — fludarabine phosphate; Mesna; Cyclophosphamide; Peripheral Blood Stem Cell Transplantation; Mycophenolic Acid; Tacrolimus; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Peripheral Blood Stem Cell Transplant (Experimental): PREPARATIVE REGIMEN: Participants receive fludarabine phosphate IV over approximately 30 minutes on days -5 to -2, and mesna IV over 24 hours and cyclophosphamide IV over approximately 2 hours on days -5 and -4. Participants also undergo total nodal irradiation on day -1.
  TRANSPLANT: Participants undergo T-Cell Receptor (TCR) alpha-beta/CD19 depleted hematopoietic stem cell transplant on day 0. If the graft contains less than 4 x 10^6 CD34+ cells/kg participant body weight (BW), patients may receive a second graft on day 1.
  GVHD PROPHYLAXIS: Participants receive mycophenolate mofetil orally twice a day (PO BID) on days -1 to 30, tacrolimus PO or IV on days 2-180 with a taper beginning on day 90 (given only if graft TCR alpha-beta+ cell content is over 1 x 10^5 cells/kg ideal BW of the patient), and rituximab IV on day 2 (given only if graft B cell content exceeds 1 x 10^5 cells/kg ideal BW of the participant).
  Interventions: Drug: Fludarabine Phosphate; Drug: Mesna; Drug: Cyclophosphamide; Radiation: Total nodal irradiation; Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation; Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Biological: Rituximab

INTERVENTIONS:
Drug: Fludarabine Phosphate — Fludarabine will be administered by IV over approximately 30 minutes for 4 days.
Drug: Mesna — Given IV over 24 hours starting prior to cyclophosphamide
Drug: Cyclophosphamide — Given IV for 2 days
Radiation: Total nodal irradiation — Undergo total lymphoid irradiation
Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation — Undergo TCR alpha-beta/DC19-depleted hematopoietic stem cell transplant
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo TCR alpha-beta/DC19-depleted hematopoietic stem cell transplant
  Other Names: HSC; HSCT
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo TCR alpha-beta/CD19-depleted hematopoietic stem cell transplant
Drug: Mycophenolate Mofetil — Given PO
  Other Names: MMF
Drug: Tacrolimus — Given PO or IV ONLY if graft cell content is over 1 x 10^5 cells/kg ideal BW of the patient
Biological: Rituximab — Given IV ONLY if graft B cell content exceeds 1 x 10^5 cells/kg ideal BW of the patient

SUMMARY:
To determine engraftment of neutrophils and platelets at 28 days following alpha/beta T-cell and CD19 cell depletion using Human Leukocyte Antigen (HLA) haploidentical donors for peripheral blood stem cell transplant in relapsed lymphoma.

Assess incidence of acute Graft Versus Host Disease (GVHD), chronic GVHD, graft failure rate, treatment related mortality rate, progression free survival and overall survival of patients.

The stem cell product will be processed using an investigational Miltenyi cell selection device/system that removes the alpha/beta T-cells and CD19+ cells, immune system cells that are more likely to cause GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet one of the following disease criteria within 24 months of registration. Salvage therapy is allowed between the participant meeting one of the below criterion and registration. Participant will be considered eligible regardless of their current disease status (i.e. complete remission, partial remission, stable disease, progressive disease) unless otherwise noted below as long as one of the below criterion has been met within the previous 24 months:

  * Relapsed/refractory Hodgkin lymphoma after autologous stem cell transplantation
  * Relapsed/refractory Hodgkin lymphoma, deemed ineligible for autologous stem cell transplantation due to refractory disease
  * Relapsed/refractory diffuse large B cell lymphoma after autologous stem cell transplantation (history of transformed lymphoma is acceptable). Disease must be in at least complete remission or partial remission with the use of salvage therapy before study treatment commences.
  * Relapsed/refractory diffuse large B cell lymphoma, deemed ineligible for autologous stem cell transplantation due to refractory disease (history of transformed lymphoma is acceptable). Disease must be in at least complete remission or partial remission with the use of salvage therapy before study treatment commences.
  * Relapsed/refractory T cell lymphoma relapsed after at least 1 prior line of therapy
  * Relapsed/refractory follicular lymphoma relapsed after at least 1 prior line of therapy
  * Relapsed/refractory mantle cell lymphoma relapsed after at least 1 prior line of therapy
  * Relapsed/refractory small lymphocytic lymphoma/chronic lymphocytic leukemia relapsed after at least 1 prior line of therapy
  * Relapsed/refractory non-Hodgkin Lymphoma, if not specified above, relapsed after at least 1 prior line of therapy
* Karnofsky score of 60% or better ("Requires occasional assistance, but is able to care for most of his/her needs").
* Pulmonary: Carbon Monoxide Diffusion Capacity (DLCO) (corrected for hemoglobin) > 40%; and Forced Expiratory Volume (FEV1) > 50%
* Cardiac: ejection fraction (EF) ≥ 50%. No uncontrolled angina or active cardiac symptoms consistent with congestive heart failure (class III or IV), by the New York Heart Association criteria. No symptomatic ventricular arrhythmias or ECG evidence of active ischemia. No evidence by echocardiography of severe valvular stenosis or regurgitation.
* Renal: estimated glomerular filtration rate (GFR) by Modification of Diet in Renal Disease (MDRD) formula > 40 mL/min/1.73m2
* Women of child bearing potential must have a negative serum or urine pregnancy test within 14 days prior to study registration and agree to use adequate birth control during study treatment. A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Voluntary written consent

Exclusion Criteria:

* Active Central nervous system (CNS) lymphoma within two weeks of registration. Patients with a history of CNS involvement must have adequate treatment as defined by at least two negative spinal fluid assessments separated by at least one week. (Otherwise Lumbar Puncture (LP) is not required if no clinical suspicion or evidence of CNS involvement.) Patients who have received cranial radiation therapy must still be eligible to receive total lymphoid irradiation to 7 Gy.
* New or active infection as determined by fever, unexplained pulmonary infiltrate or sinusitis on radiographic assessment. Infections diagnosed within 4 weeks of registration must be determined to be controlled or resolving prior to treatment.
* Presence of HIV, or active hepatitis A, B, or C infection
* Allergy or hypersensitivity to agents used within the treatment protocol.
* For an indolent lymphoma histology (follicular lymphoma, Small Lymphocytic Lymphoma/Chronic Lymphocytic Leukemia (SLL/CLL)) or mantle cell lymphoma, the patient should not have an HLA-matched sibling, who would be an eligible donor, available.
* History of prior mediastinal radiation
* Reported illicit drug use
* Vulnerable population groups, i.e., prisoners, those lacking consent capacity, non-English speaking, illiterate, pregnant females.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2021-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vaishalee P Kenkre, Principal Investigator — Principal Investigator
Locations (1):
- University of Wisconsin Carbone Cancer Center, Madison, Wisconsin, United States

REFERENCES:
- See also: UW Carbone Cancer Center Home Page — http://www.uwhealth.org/uw-carbone-cancer-center/cancer/10252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients of the University of Wisconsin Carbone Cancer Center were enrolled from March 2016 to June 2018.
Groups:
- Peripheral Blood Stem Cell Transplant: PREPARATIVE REGIMEN: Participants receive fludarabine phosphate IV over ~30 minutes on days -5 to -2, and mesna IV over 24 hours and cyclophosphamide IV over approximately 2 hours on days -5 and -4. Participants undergo total nodal irradiation on day -1.
  TRANSPLANT: Participants undergo T-Cell Receptor (TCR) alpha-beta/CD19 depleted hematopoietic stem cell transplant on day 0. If the graft contains less than 4 x 10^6 CD34+ cells/kg participant body weight (BW), Participants may receive a second graft on day 1.
  GVHD PROPHYLAXIS: Participants receive mycophenolate mofetil orally twice a day (PO BID) on days -1 to 30, tacrolimus PO or IV on days 2-180 with a taper beginning on day 90 (given only if graft TCR alpha-beta+ cell content is over 1 x 10^5 cells/kg ideal BW of the patient), and rituximab IV on day 2 (given only if graft B cell content exceeds 1 x 10^5 cells/kg ideal BW of the patient).
Period: Overall Study
Arm/Group | Peripheral Blood Stem Cell Transplant
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Peripheral Blood Stem Cell Transplant: PREPARATIVE REGIMEN: Participants receive fludarabine phosphate IV over ~30 minutes on days -5 to -2, and mesna IV over 24 hours and cyclophosphamide IV over approximately 2 hours on days -5 and -4. Participants undergo total nodal irradiation on day -1.
  TRANSPLANT: Participants undergo TCR alpha-beta/CD19 depleted hematopoietic stem cell transplant on day 0. If the graft contains less than 4 x 10^6 CD34+ cells/kg patient BW, Participants may receive a second graft on day 1.
  GVHD PROPHYLAXIS: Participants receive mycophenolate mofetil PO BID on days -1 to 30, tacrolimus PO or IV on days 2-180 with a taper beginning on day 90 (given only if graft TCR alpha-beta+ cell content is over 1 x 10^5 cells/kg ideal BW of the patient), and rituximab IV on day 2 (given only if graft B cell content exceeds 1 x 10^5 cells/kg ideal BW of the patient).
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
Age, Customized [Count of Participants; unit: Participants]
  20-29 years | 1
  30-39 years | 1
  40-49 years | 1
  50-59 years | 3
  60-69 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Absolute Neutrophil Count >= 500/Mcl for 3 Consecutive Measurements on Different Days and Platelet Count > 20,000/mm^3 With no Platelet Transfusions in the Preceding 7 Days
Description: To determine engraftment of neutrophils and platelets at 28 days following alpha/beta T-cell depletion using Human Leukocyte Antigen (HLA) haploidentical donors for stem cell transplant in relapsed lymphoma.
Time Frame: At day 28 after transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
Participants | 11

2. Secondary Outcome: Number of Participants With Grade III-IV Acute GVHD as Determined by International Bone Marrow Transplant Registry (IBMTR) Severity Index Criteria
Description: The number of participants with grade III - IV acute Graft versus host disease (GVHD) by Day +100 is reported.
Time Frame: Day +100
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
Participants | 3

3. Secondary Outcome: Number of Participants With Severe Chronic GVHD
Description: The number of participants with severe chronic GVHD by Day +180 will be reported.
Time Frame: Day +180
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
Participants | 0

4. Secondary Outcome: Number of Participants With Graft Failure
Description: Graft failure - defined as < 5% donor chimerism in the CD3 and/or CD33 selected cell populations at any time during the study follow up period once initial engraftment has been achieved.
Time Frame: Up to 2 years after graft
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
Participants | 0

5. Secondary Outcome: Number of Participants With Treatment-related Mortality
Description: Treatment-related mortality is defined as death from any cause other than disease progression.
Time Frame: Up to 2 years after graft
Measure: Count of Participants; unit: Participants
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
Participants | 4

6. Secondary Outcome: Progression-free Survival
Description: Progression-free survival will be analyzed as time before any progression by either Positron Emission Tomography/Computed Tomography (PET/CT) or bone marrow,
Time Frame: Median follow up of 1689 days
Measure: Median (Full Range); unit: days
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
days | 352 [27 to 1875]

7. Secondary Outcome: Overall Survival (OS)
Time Frame: Median follow up of 1689 days
Measure: Median (Full Range); unit: days
Arm/Group | Peripheral Blood Stem Cell Transplant
Number analyzed (Participants) | 11
days | 352 [27 to 1875]

ADVERSE EVENTS:
Time Frame: up to 5.5 years
Description: Other Adverse Events data was collected through 1 year per protocol. The data safety monitoring committee requested an additional year of data collection for serious adverse events (ie, relapses, deaths, hospitalizations, etc), SAEs are reported to 2 years per an amendment approved on 6/5/2020. All-Cause Mortality data are reported for the entire study duration, up to 5.5 years.
Arm/Group | Peripheral Blood Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 6/11
Serious Adverse Events (participants affected / at risk) | 10/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Blood Stem Cell Transplant (N=11)
Cardiac Arrest (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 3 (3)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 5 (11) — includes MRSA, Influenza A, Influenza B
Sepsis (Infections and infestations) | 2 (3)
Platelet count decreased (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Heart Failure (Cardiac disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Lung Infection (Infections and infestations) | 3 (4)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Thromboembolitic Event (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hematoma (Vascular disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Blood Bilirubin Increased (Investigations) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Death NOS (General disorders) | 1 (1)
Immune System Disorders - Other (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Peripheral Blood Stem Cell Transplant (N=11)
Abdominal pain (Gastrointestinal disorders) | 5 (12)
Acidosis (Metabolism and nutrition disorders) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (20)
Alkaline phosphatase increased (Investigations) | 4 (9)
Anemia (Blood and lymphatic system disorders) | 11 (59)
Anorexia (Metabolism and nutrition disorders) | 3 (7)
Anxiety (Psychiatric disorders) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 8 (26)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 3 (8)
Atrial flutter (Cardiac disorders) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Bloating (Gastrointestinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (10)
Blood bilirubin increased (Investigations) | 1 (2)
Blurred vision (Eye disorders) | 1 (5)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 7 (12)
Cholesterol high (Investigations) | 1 (8)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Confusion (Psychiatric disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (9)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (15)
Creatinine increased (Investigations) | 8 (24)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Delirium (Psychiatric disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 11 (33)
Dizziness (Nervous system disorders) | 6 (16)
Dry mouth (Gastrointestinal disorders) | 5 (16)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (20)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 8 (15)
Ejection fraction decreased (Investigations) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 2 (2)
Facial pain (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Fatigue (General disorders) | 9 (34)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (4)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 11 (19)
Floaters (Eye disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 2 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (4)
GGT increased (Investigations) | 3 (6)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 9 (21)
Heart failure (Cardiac disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 2 (5)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (19)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (8)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (6)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 (46)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (15)
Hypokalemia (Metabolism and nutrition disorders) | 9 (24)
Hypomagnesemia (Metabolism and nutrition disorders) | 6 (10)
Hyponatremia (Metabolism and nutrition disorders) | 7 (24)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypotension (Vascular disorders) | 6 (13)
Hypothermia (General disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (9)
Immune system disorders - Other, specify (Immune system disorders) | 4 (9)
Infections and infestations - Other, specify (Infections and infestations) | 5 (10)
INR increased (Investigations) | 3 (6)
Insomnia (Psychiatric disorders) | 5 (13)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Localized edema (General disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Lymphocyte count decreased (Investigations) | 11 (58)
Malabsorption (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 4 (6)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (5)
Multi-organ failure (General disorders) | 2 (3)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 11 (39)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neutrophil count decreased (Investigations) | 11 (29)
Non-cardiac chest pain (General disorders) | 2 (3)
Oral pain (Gastrointestinal disorders) | 3 (4)
Pain (General disorders) | 7 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (4)
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (5)
Platelet count decreased (Investigations) | 11 (59)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (7)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (3)
Proctitis (Gastrointestinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Proteinuria (Renal and urinary disorders) | 1 (4)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 (20)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (4)
Sinus tachycardia (Cardiac disorders) | 4 (9)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6 (10)
Syncope (Nervous system disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (2)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Urinary frequency (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 8 (12)
Weight loss (Investigations) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
White blood cell decreased (Investigations) | 10 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02652468/Prot_SAP_001.pdf